CLINICAL TRIAL: NCT01835249
Title: Effect of Intense vs. Standard Hypertension Management on Nighttime Blood Pressure
Brief Title: Effect of Intense vs. Standard Hypertension Management on Nighttime Blood Pressure - an Ancillary Study to SPRINT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Wake Forest University (Other); Louis Stokes VA Medical Center (U.S. Federal Agency); University of Pennsylvania (Other); Carolinas Medical Center (Other); Mayo Clinic (Other); University of Utah (Other); Vanderbilt University (Other); University of Alabama at Birmingham (Other); Michael E. DeBakey VA Medical Center (U.S. Federal Agency); Memphis VA Medical Center (U.S. Federal Agency); Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1303M30341; 1303M30341 (Other: University of Minnesota IRB)
Record Dates: First submitted 2013-04-16; First posted 2013-04-18 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Hypertension
Keywords: Hypertension; Nighttime blood pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive BP Arm (Experimental): Participants randomized into the Intensive BP arm will have a goal of SBP <120mmHg. Drugs will be added and/or titrated at each visit (monthly) to achieve SBP <120 mmHg. At periodic "milepost" visits, addition of another drug will be "required" if not at goal.
  Interventions: Other: Intensive BP Arm
- Standard BP Arm (Active Comparator): Participants randomized into the Standard arm will have a goal of SBP <140 mm Hg. Intensify therapy if SBP ≥160 mmHg @ 1 visit; ≥140 mmHg @ 2 consecutive visits; Down-titration if SBP <130 mmHg @ 1 visit; <135 mmHg @ 2 consecutive visits.
  Interventions: Other: Standard BP arm

INTERVENTIONS:
Other: Intensive BP Arm — Participants in the Intensive arm have a goal of SBP <120 mmHg.
  Arms: Intensive BP Arm
Other: Standard BP arm — Participants in the Standard BP arm have a goal of SBP <140 mmHg.
  Arms: Standard BP Arm

SUMMARY:
Hypertension is a major risk factor for cardiovascular and renal disease, and a leading cause of premature mortality worldwide. Early hypertension studies showed that treating elevated blood pressure (BP) reduces patients' risk of cardiovascular disease and all-cause mortality. In subsequent research, patients achieved greater improvement in cardiovascular outcomes when their treatment was aimed at a moderate systolic BP target (<150mmHg) than at higher targets. Although observational data suggest that even lower BP targets may be beneficial, this has not been seen in randomized trials; instead, "intense" treatment of hypertension (i.e., to a target systolic BP <120mmHg) was found to have no effect on participants' risk for renal disease, cardiovascular disease, or all-cause mortality.

One potential explanation for this apparent lack of benefit of intense BP targets is that the study protocols targeted reductions in clinic BP rather than ambulatory BP. Ambulatory BP monitoring (ABPM) allows for assessment of BP throughout the day and night. Of all the BP measurements, nighttime systolic BP appears to be the best predictor of cardiovascular disease and all-cause mortality. Because recent trials assessing intense BP targets did not include ambulatory BP measurements, the effect of intensive treatment on nighttime BP is largely unknown.

To address this important gap in knowledge, we will conduct ABPM in 600 participants as part of an ancillary study to the ongoing Systolic Blood Pressure Intervention Trial (SPRINT). The goal of the ancillary study is to evaluate the effect of intensive vs. standard clinic based BP targets on nighttime BP (primary outcome), as well as night/day BP ratio, timing of peak BP, 24hr BP, and BP variability (secondary outcomes). The SPRINT trial includes approximately 9250 participants at high risk for cardiovascular disease.

The investigators hypothesize that intense targeting of clinic systolic BP does not lower nighttime systolic BP compared to a standard target.

ELIGIBILITY:
Inclusion Criteria:

* eligible and enrolled in SPRINT at the 27 month follow up visit
* able and willing to provide informed consent

Exclusion Criteria:

* arm circumference >50cm
* shift worker or work regularly at night
* history of breast cancer requiring mastectomy
* end-stage renal disease

Min Age: 55 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 897 (Actual)
Dates: Start 2013-06; Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Nighttime systolic blood pressure | 27 month follow up visit
  Ambulatory blood pressure monitoring will be performed within 3 weeks of the 27 month follow up visit. For the primary analysis, nighttime BP will be defined by narrow clock time (01:00 AM to 6:00 AM).

SECONDARY OUTCOMES:
Night to day systolic BP ratio | 27 month follow up visit
  Ambulatory blood pressure monitoring will be performed within 3 weeks of the 27 month follow up visit. The night to day systolic BP ratio will be calculated using narrow clock times.
Timing of peak BP | 27 month follow up visit
  Ambulatory blood pressure monitoring will be performed within 3 weeks of the 27 month follow up visit. The timing of the peak BP will be calculated for each subject using cosinor rhythmometry analysis.
24hr average systolic BP | 27 month follow up visit
  Ambulatory blood pressure monitoring will be performed within 3 weeks of the 27 month follow up visit. The average systolic BP will be calculated for each subject.
Blood pressure variability | 27 month follow up visit
  Ambulatory blood pressure monitoring will be performed within 3 weeks of the 27 month follow up visit. Blood pressure variability will be defined by the standard deviation of the systolic blood pressure and by calculating the average real variability (ARV).

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Drawz, MD, MHS, MS, Principal Investigator — University of Minnesota
Locations (10):
- United States (10):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Washington DC VA Medical Center, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Florida
  - Carolinas Medical Center, Charlotte, North Carolina
  - Louis Stokes Cleveland VA Medical Center, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Memphis VA, Memphis, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Houston VA, Houston, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Result] Drawz PE, Pajewski NM, Bates JT, Bello NA, Cushman WC, Dwyer JP, Fine LJ, Goff DC Jr, Haley WE, Krousel-Wood M, McWilliams A, Rifkin DE, Slinin Y, Taylor A, Townsend R, Wall B, Wright JT, Rahman M. Effect of Intensive Versus Standard Clinic-Based Hypertension Management on Ambulatory Blood Pressure: Results From the SPRINT (Systolic Blood Pressure Intervention Trial) Ambulatory Blood Pressure Study. Hypertension. 2017 Jan;69(1):42-50. doi: 10.1161/HYPERTENSIONAHA.116.08076. Epub 2016 Nov 14. PMID 27849563